CLINICAL TRIAL: NCT06319781
Title: A Pilot Cohort Study of Risk Factors and Novel Methods of Skin Lesion Assessments in Adults With Atopic Dermatitis, Alopecia Areata, Psoriasis or Vitiligo / Et Pilot-kohortestudie om Risikofaktorer og Nye Metoder Til at Vurdere hudlæsioner Hos Voksne Med Atopisk Dermatitis, Alopecia Areata, Psoriasis Eller Vitiligo
Brief Title: A Pilot Cohort Study of Risk Factors and Novel Methods of Skin Lesion Assessments in Adults With Atopic Dermatitis, Alopecia Areata, Psoriasis or Vitiligo
Acronym: Derma-001
Status: Recruiting | Type: Observational
Sponsor: Blueskin AS (Industry)
Responsible Party: Sponsor
Other Study IDs: H-23038433
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Alopecia Areata; Vitiligo; Atopic Dermatitis; Psoriasis
MeSH Terms: conditions — Alopecia Areata; Vitiligo; Dermatitis, Atopic; Psoriasis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Atopic dermatitis: In addition to all other "basis" assessments, subjects diagnosed with AD are to complete the following forms: EASI, vIGA-AD, SCORAD, TIS, and POEM.
  Interventions: Other: Observational
- Alopecia areata: In addition to all other "basis" assessments, subjects diagnosed with AA are to complete the following forms: SALT and PGIS
  Interventions: Other: Observational
- Psoriasis: In addition to all other "basis" assessments, subjects diagnosed with psoriasis are to complete the following forms: PASI, SAPASI, PGA, PLSI
  Interventions: Other: Observational
- Vitiligo: In addition to all other "basis" assessments, subjects diagnosed with vitiligo are to complete the following forms: VASI, VETF, and VIDA
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — The study is a prospective non-interventional, observational study.

SUMMARY:
The objective of the study is to explore various clinical and biochemical parameters and their potential associations with disease severity, activity, and prognosis in atopic dermatitis, psoriasis, alopecia areata, and vitiligo. Further, the study aims at validating remote assessments of skin lesions, using smartphone-acquired photos. The study will also assess the feasibility and compliance with weekly remote-assessments and patient-reported data collection over the full study period of one year. The study will observe patients through a period of one year and will provide detailed information concerning the type and dose of medication used, as well as data to evaluate the disease activity with high resolution during this period. The study will involve collection of serum samples for exploratory biomarkers, and punch biopsies. A total of approximately 370 patients, divided into the four disease areas of atopic dermatitis, alopecia areata, psoriasis, and vitiligo, will be enrolled in the study. Using a combination of self-reported and on-site assessments and procedures, the intent is to observe the natural history of patients with select dermatological conditions, investigate tissue characteristics associated with disease activity and symptoms, and evaluate the validity of remote assessment of lesions, and feasibility of weekly self-acquired smart-phone images of skin lesions for remote assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects >18 years of age at screening.
* Previous diagnosis by a physician of atopic dermatitis, psoriasis, vitiligo, or alopecia areata.
* Visible lesions and willingness to photograph weekly using their smartphone
* Availability of a smartphone

Exclusion Criteria:

* Has any physical attributes or skin conditions that in the opinion of the investigator might interfere with the evaluation of lesions (i.e., pigmentation, tattoos, extensive scarring, excessive hair growth or acne)
* Has other clinically relevant illness that could interfere with healing of lesions (e.g. keloid scaring)
* Current or previous malignant disease, including malignant melanoma and basal cell carcinoma, within 5 years
* Some patients may have more than one of the four conditions. This is not an exclusion criterion per se but must be recorded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Minimum 18 years of age with either Atopic dermatitis, Alopecia areata, Psoriasis or Vitiligo.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Severity of the disease. | 52 weeks
  Descriptive changes in relevant disease activity scores over the study period
Clinical characteristics and disease activity. | 52 weeks
  Association/correlations of clinical characteristics (age, sex, body-mass index, baseline disease activity score, disease duration etc.) with disease activity/flares
Tissue profiling and disease activity. | 52 weeks
  Changes in tissue profiling and associations with disease activity based on relevant analyses of skin punch biopsies and standard disease activity scoring scales as listed below
Disease activity and biomarkers. | 52 weeks
  Associations of patient-reported treatment regimens and disease activity parameters, and relevant parameters derived from serum and skin biopsy biomarkers
Quality of life. | 52 weeks
  Changes from baseline in quality of life as analyzed by the WHOQOL-BREF
Compliance of remote tasks. | 52 weeks
  Proportional compliance in % with required self-assessments and photo acquisitions during the study period
Quality of smartphone collected photos. | 52 weeks
  Proportion of acquired images which were deemed of adequate quality to facilitate remote assessment
Level of agreement between the in-person and remote scoring | 52 weeks
  Level of agreement between the in-person and remote scoring, inter- and intrareliability, subsequent bias (average of differences) and precision estimates on the average difference between the scorings evaluated by the raters from remote and in-person, from the changes from baseline in relevant disease activity scores

CONTACTS AND LOCATIONS:
Overall Officials: Zarqa Ali, MD, PhD, Principal Investigator — Bispebjerg Hospital
Locations (3):
- Denmark (3):
  - Sanos Clinic, Gandrup, Gandrup
  - Sanos Clinic, Herlev, Herlev
  - Sanos Clinic, Vejle, Vejle

IPD SHARING:
Plan to Share IPD: No